CLINICAL TRIAL: NCT06846411
Title: Empagliflozin Versus Metformin for Glucose Variability and Metabolic Outcomes in Drug-Naïve Type 2 Diabetes
Brief Title: The EMPA-FIT Study
Acronym: EMPA-FIT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2201-732-003; 2021-02251 (Other Grant/Funding Number: BI)
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type II
Keywords: Metformin, empagliflozin, glucose variability
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — empagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (Active Comparator): Metformin therapy
  Interventions: Drug: Metformin
- Experimental (Experimental): Empagliflozin therapy
  Interventions: Drug: Empagliflozin 10 mg

INTERVENTIONS:
Drug: Empagliflozin 10 mg — The primary objective was to evaluate the efficacy of early treatment with empagliflozin in reducing GV, as measured by the change in MAGE from baseline to Week 12, compared to metformin.
  Arms: Experimental
Drug: Metformin — The primary objective was to evaluate the efficacy of early treatment with empagliflozin in reducing GV, as measured by the change in MAGE from baseline to Week 12, compared to metformin.
  Arms: Standard

SUMMARY:
This multicenter, open-label, prospective study randomized 46 drug-naïve adults with T2D (HbA1c 6.5%-10.0%) to receive empagliflozin (10 mg/day) or metformin (1,000 mg/day) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible if they had T2D with an HbA1c between 6.5% and 10.0%, were between 20 and 75 years of age, and had not received any anti-diabetic medications for at least eight weeks prior to screening.

Exclusion Criteria:

* individuals with a body mass index (BMI) <18.5 kg/m² or ≥40 kg/m², clinically significant hepatic impairment (e.g., hepatic cirrhosis, portal hypertension, chronic active hepatitis), or a history of acute cardiovascular events (e.g., coronary artery disease, cerebrovascular disease, peripheral arterial disease) within two months prior to enrollment. Participants with CKD (eGFR <60 mL/min/1.73 m²) or end-stage renal disease (eGFR <15 mL/min/1.73 m² or on dialysis) were also excluded.

Additional exclusion criteria included uncontrolled hypertension (BP ≥160/100 mmHg), New York Heart Association (NYHA) class III or IV heart failure, chronic oral corticosteroid use (>30 consecutive days), a history of cancer (except basal cell carcinoma) within the past five years, or significant dyslipidemia (triglycerides >1,000 mg/dL or LDL cholesterol >250 mg/dL).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
mean amplitude of glucose excursion (MAGE) | 24 weeks
  MAGE is a key glucose variability index that assesses the amplitude of clinically relevant glucose fluctuations and is calculated as the mean of the differences between consecutive glucose nadirs and peaks that exceed one standard deviation (SD) above or below the mean glucose level

SECONDARY OUTCOMES:
SD of glucose | 24 weeks
  Standard deviation of glucose obtained from continuous glucose monitoring (CGM)
Time in range (TIR) | 24 weeks
  Time in range obtained from continuous glucose monitoring (CGM)
Mean Blood Glucose (MBG) | 24 weeks
  Mean Blood Glucose (MBG) obtained from continuous glucose monitoring (CGM)
Glucose Management Indicator (GMI) | 24 weeks
  Glucose Management Indicator (GMI) obtained from continuous glucose monitoring (CGM)
Coefficient of Variation (CV) | 24 weeks
  Coefficient of Variation (CV) obtained from continuous glucose monitoring (CGM)

CONTACTS AND LOCATIONS:
Locations (1):
- SNUBH, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Anthropometric and biochemical data.
Supporting Information: Study Protocol, CSR
Time Frame: 1 year.
Access Criteria: Soo Lim